CLINICAL TRIAL: NCT00006507
Title: Occupational Therapy (OT) Outcomes: Children With Sensory Modulation Disorders
Brief Title: Occupational Therapy to Treat Children Who Over or Under React to Their Environment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NICHD-0104; 2K08 HD01183-02
Record Dates: First submitted 2000-11-04; First posted 2000-11-06 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2004-12

CONDITIONS: Sensory Disorders
Keywords: Sensory integration; Occupational therapy; Sensory Modulation Dysfunction (SMD)
MeSH Terms: conditions — Sensation Disorders | interventions — Occupational Therapy

INTERVENTIONS:
Behavioral: Occupational Therapy

SUMMARY:
Children with Sensory Modulation Dysfunction (SMD) either over- or under-react to stimuli in their environment. This can cause significant problems with daily activities and may lead to anxiety, poor attention, low self-esteem, and further complications in motor, cognitive, social and emotional development. Diagnosis of SMD is based on physiological responses to specific stimuli, measures of behavioral/social/emotional symptoms, and studies of the resulting functional limitation and disability. Treatments involve direct biomedical and behavioral intervention to improve sensory processing, as well as adjustments to the home, school and community environment. This study will compare the effect of occupational therapy vs. alternative therapy on the reactivity and function of children who have SMD.

DETAILED DESCRIPTION:
This single masked, crossover trial will randomize children with Sensory Modulation Dysfunction (SMD) to either Occupational Therapy (OT), alternative treatment (Activity Protocol), or delayed treatment (initially the control group). Children are assigned to one of the three treatment groups using a random numbers table with block randomization. Assignments are made by the research assistant, who is masked to assessments, parent priorities, and family needs/characteristics. Using block procedures, the first child is randomly assigned to treatment group A, B, or C. The next child entered to the study at that age, gender and socioeconomic status (parents' education) is randomly assigned to one of the two remaining groups. The third child meeting age, gender and SES criteria is automatically assigned to the remaining group. This procedure reduces seasonal confounds and chance variation between group characteristics. The order of treatment by group is: GROUP A (OT - 1st 10 weeks; Activity - 2nd 10 weeks); GROUP B (Activity - 1st 10 weeks; OT - 2nd 10 wks); GROUP C (Wait list - 1st 10 weeks; OT - 2nd 10 wks; Activity - 3rd 10 wks). Inclusion in the study is based on standardized assessments of physiological reactivity after a "Sensory Challenge Protocol", a technique developed by this research group and published in several medical journals. Standardized measurements of physiologic, behavioral and emotional status, are administered before treatment, after each treatment condition, and after all treatments are completed by investigators masked to treatment; and including the following:

Measurements in the Impairment: The Sensory Challenge protocol is a laboratory paradigm in which the child's physiologic reactivity after sensation is tested using electrodermal reactivity and vagal tone indices to assess sympathetic and parasympathetic systems. Measurements of functional limitations include aggression, withdrawal, impulsivity, hyperactivity, inattention, and sensitivity to tactile, movement, taste, smell, auditory and visual stimuli. These are measured in the areas: (1) attention (subscales of the parent-report Child Behavior Checklist [CBCL],and Leiter International Performance Scale-Revised; the Continuous Performance Task, the StopTask and the Go-No Go Task); (2) emotion (the CBCL); (3) sensation (the Short Sensory Profile; the Leiter-R; the Multidimensional Anxiety Scale for Children; the Stop Task; the Go-No-Go Task; the Auditory Continuous Performance Test). Measures of the Disability Dimension include the Vineland Scales of Adaptive Behavior, the Goal Attainment Scale, and play and dinner-time paradigms. Finally, measures in Societal Limitations Dimension include a parent semi-structured interview and the Visual Analogue Scale.

Occupational therapy is a targeted protocol involving functional and sensory-integration activities, supported by family-based activities at home.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sensory Modulation Disorder (children must meet all three entrance criteria): a) Physiological criteria on Sensory Challenge Protocol; b) Functional criteria on Short Sensory Profile; c) Clinical Confirmation
* IQ within normal limits (Bayley score greater than 85)

Exclusion Criteria:

* Other Diagnoses (e.g., any DSM-IV or ICD-10 diagnosed condition except ADHD)
* Previous occupational therapy
* Serious complicating life events (e.g., adoption, death of parent, abuse or neglect, foster placement, drug or alcohol exposure)
* Enrollment in Special Education or pull-out services

Ages: 54 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-03; Study Completion 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: Lucy J. Miller, Ph.D., Principal Investigator — University of Colorado Health Sciences Center, Department of Pediatrics
Locations (1):
- University of Colorado Health Sciences Center, Littleton, Colorado, United States

REFERENCES:
- [Background] Cohn E, Miller LJ, Tickle-Degnen L. Parental hopes for therapy outcomes: children with sensory modulation disorders. Am J Occup Ther. 2000 Jan-Feb;54(1):36-43. doi: 10.5014/ajot.54.1.36. PMID 10686625
- [Background] Miller, L. J., & Lane, S. J. (2000). Toward a consensus in terminology in Sensory Integration theory and practice: Part 1: Taxonomy of neurophysiological processes. Sensory Integration Special Interest Section, 23(1), 1-4.
- [Background] Ermer J, Dunn W. The sensory profile: a discriminant analysis of children with and without disabilities. Am J Occup Ther. 1998 Apr;52(4):283-90. doi: 10.5014/ajot.52.4.283. PMID 9544354
- [Background] Miller LJ, McIntosh DN, McGrath J, Shyu V, Lampe M, Taylor AK, Tassone F, Neitzel K, Stackhouse T, Hagerman RJ. Electrodermal responses to sensory stimuli in individuals with fragile X syndrome: a preliminary report. Am J Med Genet. 1999 Apr 2;83(4):268-79. PMID 10208160
- [Background] McIntosh DN, Miller LJ, Shyu V, Hagerman RJ. Sensory-modulation disruption, electrodermal responses, and functional behaviors. Dev Med Child Neurol. 1999 Sep;41(9):608-15. doi: 10.1017/s0012162299001267. PMID 10503919
- [Background] McIntosh, D.N., Miller, L.J., & Shyu, V. (1999). Overview of the Short Sensory Profile (SSP). In W. Dunn (Ed.), The sensory profile: Examiner's manual (pp. 59-83). San Antonio, TX: The Psychological Corporation.
- See also: Click here for more information about the National Institute of Child Health and Human Development. — http://www.nichd.nih.gov